CLINICAL TRIAL: NCT02794350
Title: Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Subjects (RBANS-H) in Older Patients Before and After Cochlear Implantation: A Protocol for a Prospective, Longitudinal Cohort Study
Brief Title: RBANS-H in Older Patients Before and After Cochlear Implantation: A Protocol for a Prospective Study
Acronym: RBANS-H-CI-A
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZA, Ethics Committee, University Hospital, Antwerp
Other Study IDs: 15/17/181
Record Dates: First submitted 2016-05-30; First posted 2016-06-09 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Hearing Impaired
Keywords: RBANS-H; Cochlear implantation; Cognition; Older adults; RBANS
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant

SUMMARY:
The cognitive profile of older adults with a severe to profound hearing impairment is determined by means of the Repeatable Battery for the Assessment of Neuropsychological Status, adjusted for Hearing impaired subjects (RBANS-H) before and after cochlear implantation. In this prospective, longitudinal study the participants are tested preoperatively, at six months and twelve months postoperatively and from then on yearly up to 10 years after implantation. In addition to the RBANS-H an audiological examination and an semistructured interview is conducted concerning the cochlear implant use and the self-reliance of the patient and subjective questionnaires are filled out by the subjects to assess quality of life and hearing benefit.

ELIGIBILITY:
Inclusion Criteria:

* age: 55 or older
* cochlear implant candidate (speech understanding in quiet worse than 60% at 65 decibel sound pressure level (dB SPL) in the best aided condition)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 55 or older with a severe to profound hearing loss followed-up in a tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
RBANS-H total score | Change from baseline RBANS-H total score at 6 months
  The RBANS-H assesses five cognitive domains (Immediate Memory, Visuospatial/constructional, Language, Attention and Delayed Memory). The test consists of twelve subtests and the score on each subtest contributes to one of the five domains.

SECONDARY OUTCOMES:
Best aided speech audiometry in noise: Speech reception threshold (SRT) | Change from baseline best aided SRT at 6 months
  The speech reception in noise is assessed by means of the Leuven Intelligibility Sentences Test (LIST) using an adaptive procedure. This speech material is developed to quantify the speech understanding in subjects with severely impaired hearing. The frequency spectrum of the noise signal is equal to the long-term average speech spectrum of the sentences. The level of the noise is fixed at 65 dB SPL, while the level of the speech signal is altered depending on the response of the patient. Each list consists of ten sentences and the speech reception threshold (SRT) is calculated as the mean level of the last five sentences together with the level of the imaginary 11th sentence of the list. This speech in noise test is performed both pre- and postoperatively in an aided, free field situation with the loudspeaker in front of the subject at a distance of one meter.
Nijmegen Cochlear Implant Questionnaire (NCIQ) | Change from baseline NCIQ score at 6 months
  NCIQ is a self-assessment health-related quality of life instrument developed for use in CI users. The questionnaire consists of sixty questions divided into three principal domains: Physical, Psychological and Social. The first domain comprises three subdomains, namely Basic sound perception, Advanced sound perception and Speech production. The Psychological domain contains the subdomain Self-esteem and the Social domain handles questions about Activity limitations and Social interactions. Each subdomain covers ten statements. Each statement is rated on a 5-point Likert scale ranging from 'Never' to 'Always'.
RBANS-H index scores | Change from baseline RBANS-H index scores at 6 months
  The RBANS-H assesses five cognitive domains (Immediate Memory, Visuospatial/constructional, Language, Attention and Delayed Memory). The test consists of twelve subtests and the score on each subtest contributes to one of the five domains.
Hearing thresholds: best aided Fletcher Index (FI) | Change from baseline best aided FI at 6 months
  The best-aided thresholds with hearing aid(s) and/or cochlear implant (CI) are measured through free field audiometry with warble tones. The loudspeaker is placed at a distance of one meter in front of the subject at ear level.
Speech audiometry in quiet (phoneme score): score at 65 dB SPL | Change from baseline score at 65 dB SPL at 6 months
  Speech reception in quiet is measured using Dutch open-set word lists. Each list consists of twelve monosyllabic words (consonant-vowel-consonant) of which one is a training item. One list is presented at 65 dB SPL in free field (aided, pre- and postoperatively) with a loudspeaker at 0° azimuth. The speech recognition score is the percentage of correctly identified phonemes.
Speech, Spatial and Qualities of Hearing scale 12 (SSQ12) | Change from baseline SSQ12 score at 6 months
  The SSQ12 is a short form of the Speech, Spatial and Qualities of Hearing scale. It is developed for use in clinical research and rehabilitation settings to measure a range of hearing disabilities across several domains such as speech in noise, speech in speech, localization, distance and movement, segregation and listening effort. The twelve items of this questionnaire are rated on a visual analog scale from 0 to 10 and the overall score is calculated by taking the average of the scores on these twelve items.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS score at 6 months
  To detect states of depression and anxiety the Hospital Anxiety and Depression Scale (HADS) is used. This self-assessment questionnaire consists of seven items in the subscale Depression and seven items in the subscale Anxiety and distinguishes clearly between both emotional disorders.
Hearing Implant Sound Quality Index 19 (HISQUI19) | Change from baseline HISQUI19 score at 6 months
  The HISQUI19 is a 19-item questionnaire to quantify the degree of self-perceived auditory benefit experienced by CI users in everyday communication situations. The 19 items are rated on a 7-point Likert scale ranging from always (99%) to never (1%). To calculate the overall score the corresponding numerical value of each item (from always = 7 to never = 1) is added. Uncompleted items and the response option 'not applicable' correspond to 0 in this calculation. A total score of less than 30, 30 to 59, 60 to 89, 90 to 109 and 110 to 133 is respectively classified as a very poor, poor, moderate, good and very good self-perceived auditory benefit. The validated Dutch version of the questionnaire is used.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Derived] Andries E, Bienkowska K, Swierniak W, Skarzynski PH, Skarzynski H, Calvino M, Cuadrado IS, Munoz E, Gavilan J, Lassaletta L, Tavora-Vieira D, Acharya A, Killan C, Ridgwell J, Raine C, Van de Heyning P, Van Rompaey V, Mertens G. Evolution of Type D Personality Traits After Cochlear Implantation in Severely Hearing Impaired Adults 55 Years and Older: An Exploratory Prospective, Longitudinal, Controlled, Multicenter Study. Otol Neurotol. 2022 Sep 1;43(8):e865-e871. doi: 10.1097/MAO.0000000000003622. PMID 35970164
- [Derived] Claes AJ, Mertens G, Gilles A, Hofkens-Van den Brandt A, Fransen E, Van Rompaey V, Van de Heyning P. The Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Individuals (RBANS-H) before and after Cochlear Implantation: A Protocol for a Prospective, Longitudinal Cohort Study. Front Neurosci. 2016 Nov 15;10:512. doi: 10.3389/fnins.2016.00512. eCollection 2016. PMID 27895549